CLINICAL TRIAL: NCT06369597
Title: A Randomized Controlled Trial of the Safety and Efficacy of Robotic Telesurgery Versus Laparoscopic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Robot2024
Record Dates: First submitted 2024-04-13; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Liver Cancer; Renal Cancer; Rectal Cancer
MeSH Terms: conditions — Liver Neoplasms; Kidney Neoplasms; Rectal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic telesurgery (Experimental): Patients with liver cancer, renal cancer, rectal cancer will be treated by telesurgery.
  Interventions: Procedure: Robotic telesurgery
- Laparoscopic surgery (Active Comparator): Patients with liver cancer, renal cancer, rectal cancer will be treated by laparoscopic surgery.
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Robotic telesurgery — Telesurgery by domestic surgical robot
  Arms: Robotic telesurgery
Procedure: Laparoscopic surgery — Local laparoscopic surgery
  Arms: Laparoscopic surgery

SUMMARY:
This is a randomized controlled trial that will be preceded by a safety trial focusing on the safety and efficacy of robotic telesurgery. The hypothesis is that robotic telesurgery has a non-inferior primary endpoint event rate to local laparoscopic surgery.

DETAILED DESCRIPTION:
First, a safety run-in trial for robotic telesurgery will be conducted and evaluated according to "3+3 design". At least 3 patients of each cancer type (including liver cancer,renal cancer and rectal cancer) will be enrolled for robotic telesurgery. If there is a tumor type for which the prior safety trial is terminated, the subsequent randomized controlled trial will not include patients of that type.

Second, after passing the safety run-in trial, a randomized controlled trial will be performed. New patients with each cancer type who met the enrollment criteria will be randomly assigned to either the laparoscopic surgery group(control group) or the robotic telesurgery group (intervention group) (84 patients in each group, 168 patients in total) in a 1:1 two-group parallel design.

ELIGIBILITY:
Inclusion Criteria:

* Liver Cancer:

  1. Age 18 - 75 years.
  2. Clinical diagnosis of primary hepatocellular carcinoma or benign tumor such as hepatic adenoma.
  3. Patients with hepatocellular carcinoma (BCLC stage 0-B) who were considered suitable for laparoscopic or robotic partial hepatectomy after MDT discussion, or benign tumor such as liver adenoma.
  4. ECOG score 0 ~ 1.
  5. Child-Pugh score 5 ~ 7.
* Renal cancer:

  1. Age 18 - 75 years old.
  2. Clinical diagnosis of renal cancer (cT1-T2) or benign tumor such as renal malformation tumor.
  3. Patients with benign tumors such as renal cancer (cT1-T2) or renal staggered tumor who were considered amenable to laparoscopic or robotic partial nephrectomy after MDT discussion.
  4. ECOG score 0 ~ 1.
* Rectal cancer:

  1. Age 18 - 75 years old.
  2. Clinical diagnosis of rectal cancer (Stage I-III).
  3. Patients with primary rectal cancer who are considered amenable to laparoscopic or robotic radical rectal adenocarcinoma surgery after MDT discussion.
  4. ECOG score 0 ~ 1.

Exclusion Criteria:

* Liver Cancer:

  1. Pregnant and lactating women.
  2. Combination of other malignant tumors or other malignant tumors within 5 years before enrollment.
  3. Recipients of allogeneic organ transplantation.
  4. Severe dysfunction of heart, lung, kidney and other organs.
* Renal cancer:

  1. Pregnant and lactating women.
  2. Lymph node metastasis, metastasis to other organs, previous surgical history of renal cancer, or any situation that cannot accept general anesthesia.
  3. Combination of other malignant tumors or combination of other malignant tumors within 5 years prior to enrollment.
  4. allogeneic organ transplant recipients.
  5. Severe dysfunction of heart, lungs, kidneys and other organs.
* Rectal cancer:

  1. patients with stage IV or complicated disease and emergency surgery.
  2. Pregnant and lactating women.
  3. Combination of other malignant tumors or combination of other malignant tumors within 5 years before enrollment.
  4. Allogeneic organ transplant recipients.
  5. Severe dysfunction of heart, lung, kidney and other organs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Surgical complication | One month after surgery
  Overall complication events within 30 days of surgery or intraoperative emergency intermediate open surgery events as defined by the Clavin-Dindo grading system

SECONDARY OUTCOMES:
Surgical time (min) | One month after surgery
  Total time from the start of surgery after robotic or laparoscopic installation to the end of incision closure and the surgeon's operating time.
Intraoperative blood loss (mL) | One month after surgery
  Total bleeding from the start of surgery to the end of incision suturing.
Postoperative hospitalization days | One month after surgery
  Number of days from the day of surgery to the day of discharge.
Physician satisfaction | One month after surgery
  A NASA-TLX quantification form was completed by the physician postoperatively.
Remote metrics | One month after surgery
  Record data related to network transmission end-to-end latency time, jitter, and frame loss.

CONTACTS AND LOCATIONS:
Overall Officials: Kuang Ming, PhD, Principal Investigator — First Affiliated Hospital of Sun Yat-sen University
Locations (1):
- First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No